CLINICAL TRIAL: NCT00260364
Title: A Phase I-II Dose Finding and Early Efficacy Study of Combination Therapy With Erlotinib (Tarceva), Gemcitabine, Bevacizumab (Avastin), and Capecitabine in Advanced Pancreatic Cancer
Brief Title: Combining Erlotinib Plus Bevacizumab and Gemcitabine Plus Capecitabine to Treat Advanced Pancreatic Cancer
Acronym: TARGET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Professor Cunningham's Clinical Research Fund (Unknown); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR2631; EudraCT No.: 2005-002715-24
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Cancer
Keywords: Recurrent carcinoma of the pancreas; Adenocarcinoma of the pancreas; Stage II carcinoma of the pancreas; Stage III carcinoma of the pancreas; Stage IVA carcinoma of the pancreas; Stage IVB carcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine 1000 mg/m2 iv days 1, 8, 15 of a 28 day cycle
Drug: Capecitabine orally days 1 -21
Drug: Erlotinib 100 mg orally days 1-28
Drug: Bevacizumab 5 mg/kg intravenously every 2 weeks

SUMMARY:
Pancreatic cancer is an aggressive, largely chemo-resistant disease with a poor prognosis. EGFR and VEGF are both overexpressed in pancreatic cancers and thought to contribute to tumour development and progression. The combination of gemcitabine and capecitabine has recently been shown to be effective in advanced pancreatic cancer. The combination of gemcitabine plus erlotinib has also been shown to be effective in advanced pancreatic cancer. The aim of this study is to assess whether combining a chemotherapy doublet (gemcitabine plus capecitabine) and a biologic doublet (erlotinib plus bevacizumab) is a safe and effective way to treat advanced pancreatic cancer by targeting multiple tumour stimulating mechanisms simultaneously.

DETAILED DESCRIPTION:
To establish the safety and efficacy of a combination of four drugs (capecitabine, gemcitabine, erlotinib and bevacizumab) in the treatment of patients with locally advanced or metastatic pancreatic cancer. The study will be divided into two parts:

Part A (Phase I ): Is to establish the optimal dose of capecitabine for combination with gemcitabine, bevacizumab and erlotinib. This part of the study is necessary in order to characterise any increased side effects that may occur as a result of this combination of drugs. The dose of capecitabine will be increased in cohorts containing 3 to 6 patients(according to standard dose escalation study design) whilst side effects are closely monitored. The doses of the other three drugs will remain fixed during this period:

* Gemcitabine: 1000 mg/m2 Days 1, 8, 15
* Bevacizumab: 5 mg/kg every two weeks iv
* Erlotinib: 100 mg/day orally

Maximum tolerated dose is the dose at which 2 out of a cohort of three to six patients experience dose-limiting toxicity within the first cycle (28 days) of treatment. The recommended dose for further evaluation will be one dose level below this.

Part B (Phase II): Once a recommended dose of capecitabine has been chosen, this will be used for the remainder of the trial to further characterise the efficacy and safety of the drug combination in this group of patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Locally advanced or metastatic disease
* Not amenable to curative resection
* No invasion of adjacent organs (e.g., duodenum or stomach) by CT scan
* Unidimensionally measurable disease as assessed by CT in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
* No evidence of brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin ≤ upper limit of normal
* Serum albumin > 26 g/litre

Renal:

* Creatinine ≤ 180 micromoles/litre OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular:

* No clinically significant cardiovascular disease
* No uncontrolled hypertension (i.e., blood pressure > 150/90 mm Hg on medication)
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Myocardial infarction
  * Unstable angina pectoris
  * Cerebrovascular accident
  * Transient ischemic attack
* No New York Heart Association grade II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication

OTHER:

* Not pregnant or breast feeding
* Fertile patients must use effective contraception during study participation
* No serious or non-healing wound, ulcer, or bone fracture
* No infection requiring parenteral antibiotics
* No major bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No surgery within the last 28 days or anticipation for the need for major surgery during the course of study treatment
* No other active malignancy except non-melanoma skin cancer and cervical cancer in-situ
* No history of known dihydropyrimidine dehydrogenase (DPD) deficiency
* No lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication

PRIOR CONCURRENT THERAPY:

* No previous chemotherapy, radiotherapy or other investigational drug treatment for metastatic disease (including VEGF or EGFR antagonists)
* No previous preoperative or adjuvant chemotherapy, radiotherapy or other investigational drug treatment.
* No full dose anti-coagulation (i.e. warfarin or full dose low molecular weight heparin) prior to starting study treatment.
* No ongoing treatment with aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Part A (Phase I): Dose-limiting Toxicity (DLT)
Part B (Phase II): Overall response rate (complete response and partial response)

SECONDARY OUTCOMES:
The secondary efficacy objectives of the trial are: One year survival and median overall survival
Progression free survival, Disease control rate.
The secondary safety objectives are: Toxicity,Quality of life
and Assessment of pain

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD, FRCP, Principal Investigator — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden Foundation Hospital NHS Trust, London and Surrey, London, United Kingdom